CLINICAL TRIAL: NCT05827770
Title: The Efficacy and Safety of Neoadjuvant Toripalimab Combined With Temozolomide in Resectable Stage III Melanoma: A Prospective, Single-center, Phase 2 Clinical Trial
Brief Title: The Efficacy and Safety of Neoadjuvant Toripalimab Combined With Temozolomide in Resectable Stage III Melanoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yong Chen (Other)
Responsible Party: Sponsor-Investigator, Yong Chen, Chief Physician, Fudan University
Organization: Fudan University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FU-Name-T004
Record Dates: First submitted 2023-04-09; First posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Melanoma Stage III
MeSH Terms: conditions — Melanoma | interventions — Temozolomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toripalimab Combined With Temozolomide (Experimental): Toripalimab Combined With Temozolomide
  Interventions: Drug: Toripalimab combined with Temozolomide

INTERVENTIONS:
Drug: Toripalimab combined with Temozolomide — Toripalimab combined with Temozolomide

SUMMARY:
This study is being conducted to explore the efficacy and safety of neoadjuvant toripalimab combined with temozolomide in resectable stage III melanoma.

DETAILED DESCRIPTION:
This trial is a prospective, single-center, single-arm clinical research. Unlike seen in Caucasians, checkpoint inhibitors have not obtained satisfactory results in Chinese patients. Exploring the curative effects of combination therapies in melanoma and their potential synergetic mechanism will improve the prognosis of patients. Recent retrospective data in our center showed that the objective response rate (ORR) of immunotherapy plus chemotherapy in advanced melanoma reached 40%, which was higher than immunotherapy (12.5%) and chemotherapy (4%) alone as front-line therapies. This study is aiming to evaluate the efficacy and safety of toripalimab combined with temozolomide in patients with resectable stage III melanoma. The safety and efficacy of this study will be assessed through ORR, DCR, PFS, OS, and adverse effects as graded by CTCAE 5.0.

ELIGIBILITY:
Inclusion Criteria:

* Has resectable stage IIIB-IIID melanoma of acral and cutaneous type, according to American Joint Committee on Cancer (AJCC) staging system version 8. At least one measurable lesion conforming to RECIST 1.1 criteria.
* No previously received systematic therapy of anti-PD-1 plus temozolomide. For patients with relapsed melanoma, previous therapy of anti-PD-1 plus temozolomide has been stopped for more than 6 months is acceptable.

For patients with disease progressed after receiving immune checkpoint inhibitors only, time from the last treating day is ≥ 4 weeks.

* The toxicity of prior treatment has recovered to ≤1 grade according to CTCAE 5.0.
* ECOG score 0-1.
* The expected survival time is ≥ 12 weeks.
* Adequate organ and bone marrow function.
* Female subjects of childbearing age must undergo a serum pregnancy test within 7 days before the commencement of the study and the results are negative, and are willing to use a medically approved high potency contraceptive method during the study period and within 3 months after the last administration of the study drug; For male subjects whose partner is a female of childbearing age, they should be surgically sterilized or agree to use an effective method of contraception during the study period and for 3 months after administration of the last study.
* Willing to consent and signed the informed consent, and able comply with the planned visit, research treatment, laboratory examination and other test procedures.

Exclusion Criteria:

* Has mucosal melanoma or choroidal melanoma.
* The first study drug treatment was less than 4 weeks from the last systematic antitumor therapy or 5 half-lives from the last targeted therapy; less than 4 weeks from major surgery; less than7 days from immunosuppressive drug; less than 3 weeks from immunomodulatory; less than 4 weeks from live attenuated vaccine.
* Systemic antibiotic use for 7 days within 4 weeks prior to initial administration, or unexplained fever during screening/prior to initial administration.
* With active autoimmune disease or a history of autoimmune disease.
* With history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
* With immunodeficiency, eg HIV, HBV, HCV.
* Have a clear history of serious and uncontrolled other disease or mental disorders.
* Has a bleeding tendency or abnormal clotting function.
* Known to be allergic to the active ingredients or excipients in this study.
* Other situations that the researcher considers inappropriate to participate in the research.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Pathologic response rate (pRR) | Within one week after operation
  After 2 cycles of neoadjuvant toripalimab combined with temozolomide, patients receive radical surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Yong Chen, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No